CLINICAL TRIAL: NCT04426890
Title: A Double-blind, Randomized, Active-controlled, Parallel Group, Phase 3 Study to Compare Efficacy and Safety of CT-P39 and Xolair in Patients With Chronic Spontaneous Urticaria Who Remain Symptomatic Despite H1 Antihistamine Treatment
Brief Title: To Compare Efficacy and Safety of CT-P39 and EU-approved Xolair in Patients With Chronic Spontaneous Urticaria
Acronym: omalizumab
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-P39 3.1; 2020-000952-36 (EudraCT Number)
Record Dates: First submitted 2020-06-03; First posted 2020-06-11 (Actual); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: Chronic Spontaneous Urticaria
MeSH Terms: conditions — Chronic Urticaria | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Arm 1 (Experimental): Planned to receive CT-P39 300 mg every 4 weeks in Treatment Period 1 (TP1) and maintain CT-P39 300 mg in TP2
  Interventions: Biological: CT-P39
- Arm 2 (Active Comparator): Planned to receive Xolair 300 mg every 4 weeks in TP1 and be re-randomized at Week 12 to Arm 2-1 or Arm 2-2
  Interventions: Biological: EU-approved Xolair
- Arm 2-1 (Active Comparator): Planned to receive Xolair 300 mg every 4 weeks in TP1 and be re-randomized to switch to CT-P39 300 mg in TP2
  Interventions: Biological: CT-P39; Biological: EU-approved Xolair
- Arm 2-2 (Active Comparator): Planned to receive Xolair 300 mg every 4 weeks in TP1 and be re-randomized to maintain Xolair 300 mg in TP2
  Interventions: Biological: EU-approved Xolair
- Arm 3 (Experimental): Planned to receive CT-P39 150 mg every 4 weeks in Treatment Period 1 (TP1) and increase to CT-P39 300 mg in TP2
  Interventions: Biological: CT-P39
- Arm 4 (Active Comparator): Planned to receive Xolair 150 mg every 4 weeks in Treatment Period 1 (TP1) and increase to Xolair 300 mg in TP2
  Interventions: Biological: EU-approved Xolair

INTERVENTIONS:
Biological: CT-P39 — Prefilled syringe (PFS) of 1 mL solution
  Other Names: Omalizumab
  Arms: Arm 1; Arm 2-1; Arm 3
Biological: EU-approved Xolair — Prefilled syringe (PFS) of 1 mL solution
  Other Names: Omalizumab
  Arms: Arm 2; Arm 2-1; Arm 2-2; Arm 4

SUMMARY:
A Double-blind, Randomized, Active-controlled, Parallel Group, Phase 3 Study to Compare Efficacy and Safety of CT-P39 and Xolair in Patients with Chronic Spontaneous Urticaria Who Remain Symptomatic despite H1 antihistamine Treatment

DETAILED DESCRIPTION:
CT-P39, containing the active ingredient omalizumab, is a recombinant humanized monoclonal antibody that is being developed and manufactured as a proposed biosimilar to Xolair (omalizumab) by the Sponsor. CT-P39 is identical to Xolair with respect to concentration and presentation. The 150 mg of drug product (CT-P39) will have the same pharmaceutical form and strength as 150 mg Xolair (in a prefilled syringe [PFS] for subcutaneous injection) and is intended to have a similar quality profile compared with Xolair.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with CSU
* Diagnosed as CSU refractory to H1-antihistamine

Exclusion Criteria:

* Chronic urticaria with clearly defined underlying etiology
* Clinically significant allergic reaction and/or hypersensitivity to any component of omalizumab
* History of anaphylactic shock
* History of and/or concomitant immune complex disease (including Type III hypersensitivity)
* Parasitic diseases or colonization on stool evaluation for ova and parasites
* Unable to receive background therapy with protocol-defined antihistamines or contraindicated to epinephrine

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 634 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2023-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MinJi Ma, Study Chair — Celltrion, Inc.
Locations (1):
- Klinika Ambroziak ESTEDERM, Warsaw, Poland

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 783 patients were screened for the study. Of these, 149 patients were excluded from the study due to screening failure and 634 patients were enrolled in the study. Of these 634 patients, 15 patients from the significantly GCP noncompliant study center were excluded from all analysis population. Finally, total of 619 patients were included in the data analysis.
Groups:
- Arm 1: Received CT-P39 300 mg every 4 weeks in Treatment Period 1 (TP1) and maintained CT-P39 300 mg in TP2
  CT-P39: Prefilled syringe (PFS) of 1 mL solution
- Arm 2: Received Xolair 300 mg every 4 weeks in TP1 and re-randomized at Week 12 to Arm 2-1 or Arm 2-2
  EU-approved Xolair: Prefilled syringe (PFS) of 1 mL solution
- Arm 2-1: Received Xolair 300 mg every 4 weeks in TP1 and re-randomized to switch to CT-P39 300 mg in TP2
  EU-approved Xolair: Prefilled syringe (PFS) of 1 mL solution
  CT-P39: Prefilled syringe (PFS) of 1 mL solution
- Arm 2-2: Received Xolair 300 mg every 4 weeks in TP1 and maintained Xolair 300 mg in TP2
  EU-approved Xolair: Prefilled syringe (PFS) of 1 mL solution
- Arm 3: Received CT-P39 150 mg every 4 weeks in Treatment Period 1 (TP1) and increased to CT-P39 300 mg in TP2
  CT-P39: Prefilled syringe (PFS) of 1 mL solution
- Arm 4: Received Xolair 150 mg every 4 weeks in Treatment Period 1 (TP1) and increased to Xolair 300 mg in TP2
  EU-approved Xolair: Prefilled syringe (PFS) of 1 mL solution
Period: Treatment Period 1 (Week 0 to Week 12)
Arm/Group | Arm 1 | Arm 2 | Arm 2-1 | Arm 2-2 | Arm 3 | Arm 4
Started | 204 (Among 204 patients, one patient in Arm 1 who was randomized by mistake terminated the study prior to the first study drug administration.) | 205 | 0 | 0 | 107 | 103
Completed (Refers Study drug completion) | 187 | 192 | 0 | 0 | 101 | 98
Not Completed | 17 | 13 | 0 | 0 | 6 | 5
Period: Treatment Period 2 (Week 12 to Week 24)
Arm/Group | Arm 1 | Arm 2 | Arm 2-1 | Arm 2-2 | Arm 3 | Arm 4
Started (Only patients who entered into TP2 and were administered with assigned study drug in TP2 are included.) | 187 | 0 | 96 | 96 | 101 | 98
Completed (Refers Study drug completion) | 181 | 0 | 94 | 94 | 99 | 94
Not Completed | 6 | 0 | 2 | 2 | 2 | 4
Period: Follow Up Period
Arm/Group | Arm 1 | Arm 2 | Arm 2-1 | Arm 2-2 | Arm 3 | Arm 4
Started (All patients who entered into Follow up period are included regardless of study drug completion) | 182 | 184 (Of these, two patients were not re-randomized in the TP2 (not initiated the TP2), and entered into the follow-up period.) | 0 (Total of 90 patients assigned in Arm 2-1 in TP2 entered into follow-up period.) | 0 (Total of 92 patients assigned in Arm 2-2 in TP2 entered into follow-up period.) | 98 | 90
Completed | 172 | 172 | 0 (Among 90 patients, 84 patients completed follow-up period.) | 0 (Among 92 patients, 86 patients completed follow-up period.) | 91 | 83
Not Completed | 10 | 12 | 0 | 0 | 7 | 7

BASELINE CHARACTERISTICS:
Population: The RAN Set was defined as all randomly assigned patients prior to dosing on Day 1 regardless of whether they received any study drug (CT-P39 or Xolair).
Groups:
- Arm 1: Received 300 mg of CT-P39 as SC injections via PFS during Treatment Period (TP1)
  CT-P39: Prefilled syringe (PFS) of 1 mL solution
- Arm 2: Received 300 mg of EU-approved Xolair as SC injections via PFS during TP1
  EU-approved Xolair: Prefilled syringe (PFS) of 1 mL solution
- Arm 3: Received 150 mg of CT-P39 as SC injections via PFS during TP1
  CT-P39: Prefilled syringe (PFS) of 1 mL solution
- Arm 4: Received 150 mg of EU-approved Xolair as SC injections via PFS during TP1
  EU-approved Xolair: Prefilled syringe (PFS) of 1 mL solution
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Total
Number analyzed (Participants) | 204 | 205 | 107 | 103 | 619
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (13.3) | 42.9 (13.7) | 42.9 (15.0) | 41.5 (13.8) | 42.8 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 131 | 67 | 72 | 403
  Male | 71 | 74 | 40 | 31 | 216
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 38 | 40 | 21 | 20 | 119
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 166 | 165 | 86 | 83 | 500
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Bulgaria | 40 | 42 | 23 | 20 | 125
  Greece | 3 | 1 | 1 | 1 | 6
  Hungary | 1 | 2 | 2 | 1 | 6
  South Korea | 38 | 40 | 21 | 20 | 119
  Poland | 87 | 87 | 43 | 45 | 262
  Ukraine | 35 | 33 | 17 | 16 | 101
Baseline ISS7 [Count of Participants; unit: Participants] — The ISS was recorded twice daily (morning and evening) in the patient eDiary, on scale of 0 (none) to 3 (severe) points. The daily ISS is the average of the morning and evening scores and the ISS7 is the sum of the daily ISS over 7 days. The baseline ISS7 is the sum of the daily ISS over the 7 days (Day -7 to -1) prior to the first study drug administration. The ISS7 can range from 0 to 21. The higher scores mean a worse outcome.
  Participants
    < 13 points | 36 | 42 | 20 | 17 | 115
    ≥ 13 points | 168 | 163 | 87 | 86 | 504
Weight on Day 1, [Count of Participants; unit: Participants]
  < 80 kg | 123 | 125 | 65 | 65 | 378
  ≥ 80 kg | 81 | 80 | 42 | 38 | 241

OUTCOME MEASURES:

1. Primary Outcome: Therapeutic Equivalence Based on Change From Baseline in ISS7 at Week 12 in 300 mg Groups
Description: The primary efficacy evaluation was comparison of mean change from baseline in ISS7 of 300 mg of CT-P39 (Arm 1) and 300 mg of Xolair (Arm 2) at Week 12, calculated as ISS7 at Week 12 minus the baseline ISS7. The ISS was recorded twice daily (morning and evening) in the patient eDiary, on scale of 0 (none) to 3 (severe) points. The daily ISS is the average of the morning and evening scores and the ISS7 is the sum of the daily ISS over 7 days. The ISS7 can range from 0 to 21. The higher scores mean a worse outcome.
  The analysis was conducted by analysis of covariance (ANCOVA). The ANCOVA model included the treatment group as a fixed effect and baseline ISS7, body weight on Day 1 and country as covariates.
Time Frame: Week 12
Population: Analysis was performed based on mITT Set which had different definition with RAN set for disposition table.
  This table presents the actual number of patients who had a result and were included in the analysis.
  The mITT Set was defined as all randomly assigned patients who received at least 1 full dose of either of the study drugs during Treatment Period I.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Arm 1: Received 300 mg of CT-P39 as SC injections via PFS during Treatment Period 1 (TP1)
  CT-P39: Prefilled syringe (PFS) of 1 mL solution
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 203 | 205
score on a scale | -9.25 (0.787) | -9.96 (0.791)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; The statistical analysis of mean change from baseline in ISS7 at Week 12 between CT-P39 300 mg treatment arm (Arm 1) and Xolair 300 mg treatment arm (Arm 2), using ANCOVA with multiple imputation based on the MAR assumption was performed for the mITT Set; Test type: Equivalence — Therapeutic equivalence was declared if the two-sided 90% confidence interval (CI) for the treatment difference was entirely within an equivalence margin of [-2.5, 2.0]; Mean Difference (Net) = 0.70, 90% CI 2-sided [-0.22 to 1.63]

2. Primary Outcome: Relative Potency of CT-P39 Compared With Xolair Based on Change From Baseline in ISS7 at Week 12
Description: The ISS was recorded twice daily (morning and evening) in the patient eDiary, on scale of 0 (none) to 3 (severe) points. The daily ISS is the average of the morning and evening scores and the ISS7 is the sum of the daily ISS over 7 days. The ISS7 can range from 0 to 21. The higher scores mean a worse outcome.
  The relative potency was not calculated due to the assumption of parallel-line assay not being met. A parallel-line assay assumes that dose-efficacy response relationships are linear and parallel on log-dose scale which requires the equal slope in the regression model used to estimate relative potency. However, the slopes of the two treatment groups were estimated to be different, indicating a violation of the parallelism assumption. As a result, the relative potency was not computed.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: participants
Groups:
- Arm 3: Received 150mg of CT-P39 as SC injections via PFS during TP1
  CT-P39: Prefilled syringe (PFS) of 1 mL solution
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 203 | 205 | 107 | 103
participants | NA [NA to NA] — The relative potency was not calculated due to assumption of parallel-line assay not being met. | NA [NA to NA] — The relative potency was not calculated due to assumption of parallel-line assay not being met. | NA [NA to NA] — The relative potency was not calculated due to assumption of parallel-line assay not being met. | NA [NA to NA] — The relative potency was not calculated due to assumption of parallel-line assay not being met.

3. Secondary Outcome: Change From Baseline in Weekly Itch Severity Score (ISS7) at Week 12
Description: The change from baseline in ISS7 at Week 12 was calculated as ISS7 at Week 12 minus the baseline ISS7. The ISS was recorded twice daily (morning and evening) in the patient eDiary, on scale of 0 (none) to 3 (severe) points. The daily ISS is the average of the morning and evening scores and the ISS7 is the sum of the daily ISS over 7 days. The ISS7 can range from 0 to 21. The higher scores mean a worse outcome. The relative potency based on the CFB of ISS7 at Week 12 was not calculated due to assumption of parallel-line assay not being met.
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 186 | 192 | 101 | 94
score on a scale | -9.31 (6.20) | -9.99 (6.18) | -9.56 (5.87) | -8.73 (6.65)

4. Secondary Outcome: Change From Baseline in Weekly Itch Severity Score (ISS7) at Week 24
Description: The change from baseline in ISS7 at Week 24 was calculated as ISS7 at Week 24 minus the baseline ISS7. The ISS was recorded twice daily (morning and evening) in the patient eDiary, on scale of 0 (none) to 3 (severe) points. The daily ISS is the average of the morning and evening scores and the ISS7 is the sum of the daily ISS over 7 days. The ISS7 can range from 0 to 21. The higher scores mean a worse outcome.
Time Frame: Week 24
Population: Analysis was performed based on mITT-TP2 Subset which had different definition with RAN set for disposition table.
  This table presents the actual number of patients who had a result and were included in the analysis.
  The mITT-TP2 Subset was defined as all patients in the mITT Set who underwent the second randomization and received at least 1 full dose of either of the study drugs during Treatment Period II.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Arm 1: Received CT-P39 300 mg in Treatment Period 1 (TP1) and maintained CT-P39 300 mg in Treatment Period 2 (TP2)
  CT-P39: Prefilled syringe (PFS) of 1 mL solution
- Arm 2-1: Received Xolair 300 mg in TP1 and switched to CT-P39 300 mg in TP2
  CT-P39: Prefilled syringe (PFS) of 1 mL solution
  EU-approved Xolair: Prefilled syringe (PFS) of 1 mL solution
- Arm 2-2: Received Xolair 300 mg in TP1 and maintained Xolair 300 mg in TP2
  EU-approved Xolair: Prefilled syringe (PFS) of 1 mL solution
- Arm 3: Received CT-P39 150 mg in TP1 and increased to CT-P39 300 mg in TP2
  CT-P39: Prefilled syringe (PFS) of 1 mL solution
- Arm 4: Received Xolair 150 mg in TP1 and increased to Xolair 300 mg in TP2
  EU-approved Xolair: Prefilled syringe (PFS) of 1 mL solution
Arm/Group | Arm 1 | Arm 2-1 | Arm 2-2 | Arm 3 | Arm 4
Number analyzed (Participants) | 170 | 88 | 82 | 90 | 86
score on a scale | -11.22 (6.21) | -12.24 (5.69) | -11.19 (5.88) | -11.76 (5.61) | -10.70 (6.17)

5. Secondary Outcome: Time to Minimally Important Difference (MID) in ISS7 by Week 12
Description: Time to MID response was the time (in weeks) from Day 1 to the study week when reduction of 5 points or more from baseline for ISS7 was first achieved up to Week 12. If a patient failed to achieve an MID response up to Week 12 or terminated the study prior to Week 12 without achieving MID response, the patient was censored at the date (in weeks) of the last non-missing ISS7 evaluation. Time to MID was estimated by Kaplan-Meier method. The lower result means a better outcome.
Time Frame: Up to Week 12
Population: Analysis was performed based on mITT Set which had different definition with RAN set for disposition table.
  The mITT Set was defined as all randomly assigned patients who received at least 1 full dose of either of the study drugs during Treatment Period I.
Measure: Median (95% Confidence Interval); unit: in Weeks
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 203 | 205 | 107 | 103
in Weeks | 2.00 [2.00 to 3.00] | 2.00 [2.00 to 3.00] | 2.00 [2.00 to 3.00] | 2.00 [2.00 to 3.00]

6. Secondary Outcome: Percentage of Minimally Important Difference (MID) Responders in ISS7 at Week 12
Description: Number of patients who achieved MID response at Week 12 were presented. MID response is a change from baseline in ISS7 of ≤ -5. If a patient had missing weekly scores for the given week the patient was classified as a non-responder. The higher percentage means a better outcome.
Time Frame: Week 12
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 203 | 205 | 107 | 103
Participants | 141 | 152 | 78 | 65

7. Secondary Outcome: Change From Baseline in Weekly Hives Severity Score (HSS7) at Week 12
Description: The change from baseline in HSS7 at Week 12 was calculated as HSS7 at Week 12 minus the baseline HSS7. The HSS was counted twice daily (morning and evening) in the patient eDiary, on a scale of 0 (none) to 3 (intense) points. The daily HSS is the average of the morning and evening scores, and the HSS7 is the sum of the daily HSS over 7 days. HSS7 can range from 0 to 21. The higher scores mean a worse outcome.
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 186 | 192 | 101 | 94
score on a scale | -9.96 (6.88) | -10.55 (6.93) | -10.29 (6.75) | -9.48 (6.93)

8. Secondary Outcome: Change From Baseline in Weekly Hives Severity Score (HSS7) at Week 24
Description: The change from baseline in HSS7 at Week 24 was calculated as HSS7 at Week 24 minus the baseline HSS7. The HSS was counted twice daily (morning and evening) in the patient eDiary, on a scale of 0 (none) to 3 (intense) points. The daily HSS is the average of the morning and evening scores, and the HSS7 is the sum of the daily HSS over 7 days. HSS7 can range from 0 to 21. The higher scores mean a worse outcome.
Time Frame: Week 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 | Arm 2-1 | Arm 2-2 | Arm 3 | Arm 4
Number analyzed (Participants) | 170 | 88 | 82 | 90 | 86
score on a scale | -11.86 (6.72) | -12.72 (6.72) | -12.36 (6.64) | -12.74 (6.01) | -11.77 (6.20)

9. Secondary Outcome: Change From Baseline in Weekly Urticaria Activity Score (UAS7) at Week 12
Description: The change from baseline in UAS7 at Week 12 was calculated as UAS7 at Week 12 minus the baseline UAS7. The UAS was calculated as the sum of the ISS and the HSS by diary-based documentation. The sum of the scores represented disease severity on a scale from 0 (minimum) to 6 (maximum). The daily UAS is the average of the morning and evening scores and the UAS7 is the sum of the daily UAS over 7 days. UAS7 can range from 0 to 42. The higher scores mean a worse outcome.
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 186 | 192 | 101 | 94
score on a scale | -19.27 (12.53) | -20.54 (12.69) | -19.84 (12.02) | -18.21 (13.06)

10. Secondary Outcome: Change From Baseline in Weekly Urticaria Activity Score (UAS7) at Week 24
Description: The change from baseline in UAS7 at Week 24 was calculated as UAS7 at Week 24 minus the baseline UAS7. The UAS was calculated as the sum of the ISS and the HSS by diary-based documentation. The sum of the scores represented disease severity on a scale from 0 (minimum) to 6 (maximum). The daily UAS is the average of the morning and evening scores and the UAS7 is the sum of the daily UAS over 7 days. UAS7 can range from 0 to 42. The higher scores mean a worse outcome.
Time Frame: Week 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 | Arm 2-1 | Arm 2-2 | Arm 3 | Arm 4
Number analyzed (Participants) | 170 | 88 | 82 | 90 | 86
score on a scale | -23.08 (12.30) | -24.96 (11.79) | -23.55 (12.08) | -24.50 (11.13) | -22.48 (11.84)

11. Secondary Outcome: Percentage of Patients With UAS7 of ≤ 6 Points and Complete Responders in Weekly Urticaria Activity Score at Week 12
Description: Percentage of patients with Weekly Urticaria Activity Score (UAS7) of ≤ 6 points and complete responders (UAS7 = 0) at Week 12 is presented. If a patient had missing weekly scores for the given week the patient was classified as a non-responder. UAS7 can range from 0 to 42. The higher result means a better outcome.
Time Frame: Week 12
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 203 | 205 | 107 | 103
Participants
  Patients with UAS7 ≤ 6 | 77 | 83 | 41 | 33
  Patients with UAS7 = 0 | 48 | 63 | 23 | 14

12. Secondary Outcome: Percentage of Patients With UAS7 of ≤ 6 Points and Complete Responders in Weekly Urticaria Activity Score at Week 24
Description: The number of patients with Weekly Urticaria Activity Score (UAS7) of ≤ 6 points and complete responders (UAS7 = 0) at Week 24 is presented. If a patient had missing weekly scores for the given week the patient was classified as a non-responder. UAS7 can range from 0 to 42. The higher result means a better outcome.
Time Frame: Week 24
Population: Analysis was performed based on mITT-TP2 Subset which had different definition with RAN set for disposition table.
  The mITT-TP2 Subset was defined as all patients in the mITT Set who underwent the second randomization and received at least 1 full dose of either of the study drugs during Treatment Period II.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2-1 | Arm 2-2 | Arm 3 | Arm 4
Number analyzed (Participants) | 187 | 96 | 96 | 101 | 98
Participants
  Patients with UAS7 of ≤ 6 | 102 | 65 | 46 | 55 | 41
  Patients with UAS7 = 0 | 75 | 49 | 36 | 39 | 31

13. Secondary Outcome: Percentage of Angioedema-Free Days From Week 4 to Week 12
Description: The proportion of angioedema-free days from Week 4 to Week 12 is defined as the number of days for which the patient indicated a 'No' response to the angioedema question in the patient eDiary divided by the total number of days with a non-missing diary entry starting on Week 4 visit date and ending the day prior to Week 12 visit date. Patients who had missing responses for > 40% of the daily diary entries between Week 4 visit date and Week 12 visit date were not included in this analysis. The higher result means a better outcome.
Time Frame: Week 4 to 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of Angioedema-Free Days
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 189 | 190 | 99 | 97
percentage of Angioedema-Free Days | 93.47 (17.95) | 90.14 (25.64) | 96.94 (10.83) | 93.77 (18.01)

14. Secondary Outcome: Change From Baseline in Number of Tablets/Week of Rescue Therapy at Week 12
Description: The change from baseline in the number of tablets/week of rescue therapy used at Week 12 is presented. The number of tablets for each week of rescue therapy will be defined as the sum of daily use of rescue therapy over the study days which make up a given study week. The higher value means a worse outcome.
  If a subject switched rescue therapy medication and started a different medication or the prescribed dose of the rescue therapy medication changed during the study, the subject was excluded from the summary.
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of Tablets/Week
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 170 | 180 | 92 | 85
Number of Tablets/Week | -1.33 (3.73) | -1.45 (3.16) | -1.19 (2.71) | -1.53 (3.42)

15. Secondary Outcome: Change From Baseline in Number of Tablets/Week of Rescue Therapy at Week 24
Description: The change from baseline in the number of tablets/week of rescue therapy used at Week 24 is presented. The number of tablets for each week of rescue therapy will be defined as the sum of daily use of rescue therapy over the study days which make up a given study week. The higher value means a worse outcome.
  If a subject switched rescue therapy medication and started a different medication or the prescribed dose of the rescue therapy medication changed during the study, the subject was excluded from the summary.
Time Frame: Week 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Number of Tablets/Week
Arm/Group | Arm 1 | Arm 2-1 | Arm 2-2 | Arm 3 | Arm 4
Number analyzed (Participants) | 154 | 78 | 79 | 81 | 78
Number of Tablets/Week | -1.40 (3.79) | -1.75 (3.67) | -1.74 (2.98) | -1.50 (3.36) | -1.77 (3.33)

16. Secondary Outcome: Change From Baseline in the Overall Dermatology Life Quality Index (DLQI) Score at Week 12
Description: The change from baseline in mean overall DLQI score at Week 12 is presented. The DLQI is a 10-item dermatology-specific health-related questionnaire across 6 domains: symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. Patients rated their dermatology symptoms as well as the impact of their skin condition on various aspect of their lives. Each question is scored from 0 to 3. Overall DLQI ranges on a scale of 0 to 30. The higher result means a worse outcome.
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 169 | 179 | 98 | 91
score on a scale | -8.9 (7.5) | -9.0 (6.7) | -9.2 (7.0) | -8.9 (8.2)

17. Secondary Outcome: Change From Baseline in the Overall Dermatology Life Quality Index (DLQI) Score at Week 24
Description: The change from baseline in mean overall DLQI score at Week 24 is presented. The DLQI is a 10-item dermatology-specific health-related questionnaire across 6 domains: symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. Patients rated their dermatology symptoms as well as the impact of their skin condition on various aspect of their lives. Each question is scored from 0 to 3. Overall DLQI ranges on a scale of 0 to 30. The higher result means a worse outcome.
Time Frame: Week 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 | Arm 2-1 | Arm 2-2 | Arm 3 | Arm 4
Number analyzed (Participants) | 161 | 87 | 87 | 93 | 89
score on a scale | -9.4 (6.9) | -10.4 (7.3) | -9.8 (6.9) | -10.5 (7.7) | -10.1 (7.5)

18. Secondary Outcome: Change From Baseline in the Overall Chronic Urticaria Quality of Life Questionnaire Score (CU-Q2oL) Score at Week 12
Description: The change from baseline in mean overall CU-Q2oL score at Week 12 is presented. The CU-Q2oL is a 23-item CSU specific health-related QoL questionnaire across 6 domains: pruritus, swelling, impact on life activities, sleep problems, limits, and looks. Patients rated their CSU symptoms and the impact of their CSU on various aspects of their lives. Each question was scored from 1 (not at all) to 5 (extremely), and overall raw score, on a scale of 23 to 115, was calculated by summing the individual raw domain scores. The higher result means a worse outcome.
  Overall raw scores of CU-Q2oL were converted to 0 to 100 point scores according to the following formula:[(sum of items - minimum) / (maximum - minimum)] × 100, where minimum=23 (1 score for all 23 items), maximum=115 (5 score for all 23 items).
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 178 | 186 | 100 | 94
score on a scale | -25.40 (20.33) | -28.11 (19.93) | -27.32 (20.81) | -26.51 (23.27)

19. Secondary Outcome: Change From Baseline in the Overall Chronic Urticaria Quality of Life Questionnaire Score (CU-Q2oL) Score at Week 24
Description: The change from baseline in mean overall CU-Q2oL score at Week 24 is presented. The CU-Q2oL is a 23-item CSU specific health-related QoL questionnaire across 6 domains: pruritus, swelling, impact on life activities, sleep problems, limits, and looks. Patients rated their CSU symptoms and the impact of their CSU on various aspects of their lives. Each question was scored from 1 (not at all) to 5 (extremely), and overall raw score, on a scale of 23 to 115, was calculated by summing the individual raw domain scores. The higher result means a worse outcome.
  Overall raw scores of CU-Q2oL were converted to 0 to 100 point scores according to the following formula: [(sum of items - minimum) / (maximum - minimum)] × 100, where minimum=23 (1 score for all 23 items), maximum=115 (5 score for all 23 items)
Time Frame: Week 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 | Arm 2-1 | Arm 2-2 | Arm 3 | Arm 4
Number analyzed (Participants) | 167 | 90 | 89 | 94 | 90
score on a scale | -29.19 (18.76) | -31.33 (21.95) | -31.88 (22.33) | -31.71 (19.96) | -30.88 (22.22)

20. Secondary Outcome: Trough Serum Concentration (Ctrough) of Omalizumab at Week 12
Description: All concentration below lower limit of quantification (BLQ) values were treated as zero (0) for PK parameter summary. Below lower limit of quantification (BLQ) is treated as zero (0).
Time Frame: Week 12
Population: Analysis was performed based on PK Set which had different definition with RAN set for disposition table.
  This table presents the actual number of patients who had a result and were included in the analysis.
  The PK Set was defined as all patients who received at least 1 full dose of either of the study drugs during Treatment Period I and had at least 1 post-treatment PK result prior to dosing at Week 12.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 187 | 193 | 101 | 97
ug/mL | 31.50791 (12.11966) | 31.35679 (13.44334) | 14.67465 (6.31588) | 15.80010 (7.65671)

21. Secondary Outcome: Trough Serum Concentration (Ctrough) of Omalizumab at Week 24
Description: as for outcome 20
Time Frame: Week 24
Population: Analysis was performed based on PK-TP2 Subset which had different definition with RAN set for disposition table.
  This table presents the actual number of patients who had a result and were included in the analysis.
  The PK-TP2 Subset was defined as all patients in PK Set who received at least 1 full dose of either of the study drugs during Treatment Period II and had at least 1 post-treatment PK result after Week 12
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Arm 1 | Arm 2-1 | Arm 2-2 | Arm 3 | Arm 4
Number analyzed (Participants) | 177 | 92 | 94 | 97 | 92
ug/mL | 35.43099 (14.98897) | 35.87102 (18.09287) | 33.50606 (14.25536) | 30.41523 (13.16691) | 33.63630 (16.55088)

22. Secondary Outcome: Immunogenicity Result at Week 12
Description: Anti-drug Antibody test involved both screening and confirmatory assays to confirm true positive results. Samples that are positive in the screening assay underwent further testing in the confirmatory assay to determine if patients are true positive. Samples that are positive in the ADA confirmatory assay were analyzed further to conduct a NAb assessment.
Time Frame: Week 12
Population: Analysis was performed based on Safety Set which had different definition with RAN set for disposition table.
  This table presents the actual number of patients who had a result and were included in the analysis.
  The Safety Set was defined as all randomly assigned patients who received at least 1 dose (full or partial) of either of the study drugs.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 203 | 205 | 107 | 103
Participants
  ADA positive | 1 | 0 | 2 | 0
  NAb positive (in ADA positive patients) | 1 | 0 | 1 | 0

23. Secondary Outcome: Immunogenicity Result at Week 24
Description: as for outcome 22
Time Frame: Week 24
Population: Analysis was performed based on Safety-TP2 Subset which had different definition with RAN set for disposition table.
  This table presents the actual number of patients who had a result and were included in the analysis.
  The Safety-TP2 Subset was defined as all patients in Safety Set who received at least 1 dose (full or partial) of either of the study drugs during Treatment Period II.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2-1 | Arm 2-2 | Arm 3 | Arm 4
Number analyzed (Participants) | 187 | 96 | 96 | 101 | 98
Participants
  ADA positive | 9 | 2 | 0 | 4 | 1
  NAb positive (in ADA positive patients) | 2 | 0 | 0 | 3 | 1

ADVERSE EVENTS:
Time Frame: Treatment-Emergent Adverse Event Up to Week 40. The 'Other Adverse Events' table includes only non-serious treatment-emergent AEs that occurred in ≥2% of patients in at least one arm/period group. Each patient is counted only once, even if they reported multiple AEs for the total patient number of each arm/period group.
Description: The data includes treatment-emergent adverse event during overall period. For treatment Period 2, the summary is presented in the Safety TP2 Subset, and Others are presented in the Safety Set.
  The Safety Set was defined as all randomly assigned patients who received at least 1 dose (full or partial) of either of the study drugs.
  The Safety-TP2 Subset was defined as all patients in Safety Set who received at least 1 dose (full or partial) of either of the study drugs during Treatment Period II.
Groups:
- Arm 1/Treatment Period 1; Arm 1/Follow-up Period: Received 300 mg of CT-P39 as SC injections via PFS in Treatment Period 1 (TP1)
  CT-P39: Prefilled syringe (PFS) of 1 mL solution
- Arm 2/ Treatment Period 1; Arm 2/Follow-up Period: Received 300 mg of EU-approved Xolair as SC injections via PFS in TP1
  EU-approved Xolair: Prefilled syringe (PFS) of 1 mL solution
- Arm 3/ Treatment Period 1; Arm 3/Follow-up Period: Received 150mg of CT-P39 as SC injections via PFS in TP1
  CT-P39: Prefilled syringe (PFS) of 1 mL solution
- Arm 4/ Treatment Period 1; Arm 4/Follow-up Period: Received 150 mg of EU-approved Xolair as SC injections via PFS in TP1
  EU-approved Xolair: Prefilled syringe (PFS) of 1 mL solution
- Arm 1/Treatment Period 2: Received 300 mg of CT-P39 as SC injections via PFS in Treatment Period 1 (TP1) and maintained CT-P39 300 mg in Treatment Period 2 (TP2)
  CT-P39: Prefilled syringe (PFS) of 1 mL solution
- Arm 2-1/ Treatment Period 2: Received 300 mg of EU-approved Xolair as SC injection via PFS in TP1 and switched to CT-P39 300 mg in TP2
  CT-P39: Prefilled syringe (PFS) of 1 mL solution
  EU-approved Xolair: Prefilled syringe (PFS) of 1 mL solution
- Arm 2-2/Treatment Period 2: Received 300 mg of EU-approved Xolair as SC injection via PFS in TP1 and maintained Xolair 300 mg in TP2
  EU-approved Xolair: Prefilled syringe (PFS) of 1 mL solution
- Arm 3/ Treatment Period 2: Received 150 mg of CT-P39 as SC injections via PFS in TP1 and increased to CT-P39 300 mg in TP2
  CT-P39: Prefilled syringe (PFS) of 1 mL solution
- Arm 4/ Treatment Period 2: Received 150 mg of EU-approved Xolair as SC injections via PFS in TP1 and increased to Xolair 300 mg in TP2
  EU-approved Xolair: Prefilled syringe (PFS) of 1 mL solution
Arm/Group | Arm 1/Treatment Period 1 | Arm 2/ Treatment Period 1 | Arm 3/ Treatment Period 1 | Arm 4/ Treatment Period 1 | Arm 1/Treatment Period 2 | Arm 2-1/ Treatment Period 2 | Arm 2-2/Treatment Period 2 | Arm 3/ Treatment Period 2 | Arm 4/ Treatment Period 2 | Arm 1/Follow-up Period | Arm 2/Follow-up Period | Arm 3/Follow-up Period | Arm 4/Follow-up Period
All-Cause Mortality (participants affected / at risk) | 0/203 | 0/205 | 0/107 | 0/103 | 1/187 | 0/96 | 0/96 | 0/101 | 0/98 | 0/203 | 0/205 | 0/107 | 0/103
Serious Adverse Events (participants affected / at risk) | 4/203 | 2/205 | 2/107 | 3/103 | 5/187 | 0/96 | 2/96 | 0/101 | 0/98 | 1/203 | 4/205 | 3/107 | 0/103
Other Adverse Events (participants affected / at risk) | 22/203 | 23/205 | 16/107 | 12/103 | 16/187 | 8/96 | 10/96 | 8/101 | 5/98 | 8/203 | 17/205 | 8/107 | 7/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1/Treatment Period 1 (N=203) | Arm 2/ Treatment Period 1 (N=205) | Arm 3/ Treatment Period 1 (N=107) | Arm 4/ Treatment Period 1 (N=103) | Arm 1/Treatment Period 2 (N=187) | Arm 2-1/ Treatment Period 2 (N=96) | Arm 2-2/Treatment Period 2 (N=96) | Arm 3/ Treatment Period 2 (N=101) | Arm 4/ Treatment Period 2 (N=98) | Arm 1/Follow-up Period (N=203) | Arm 2/Follow-up Period (N=205) | Arm 3/Follow-up Period (N=107) | Arm 4/Follow-up Period (N=103)
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femoral hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronavirus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tryptase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Behcet's syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chronic Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1/Treatment Period 1 (N=203) | Arm 2/ Treatment Period 1 (N=205) | Arm 3/ Treatment Period 1 (N=107) | Arm 4/ Treatment Period 1 (N=103) | Arm 1/Treatment Period 2 (N=187) | Arm 2-1/ Treatment Period 2 (N=96) | Arm 2-2/Treatment Period 2 (N=96) | Arm 3/ Treatment Period 2 (N=101) | Arm 4/ Treatment Period 2 (N=98) | Arm 1/Follow-up Period (N=203) | Arm 2/Follow-up Period (N=205) | Arm 3/Follow-up Period (N=107) | Arm 4/Follow-up Period (N=103)
COVID-19 (Infections and infestations) | 5 | 7 | 4 | 1 | 5 | 2 | 1 | 2 | 3 | 2 | 8 | 4 | 5
Dizziness (Nervous system disorders) | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 5 | 5 | 0 | 4 | 1 | 1 | 2 | 0 | 1 | 2 | 0 | 3 | 1
Immunisation reaction (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 5 | 9 | 1 | 3 | 1 | 3 | 2 | 1 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 7 | 4 | 7 | 2 | 6 | 2 | 4 | 1 | 0 | 3 | 7 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 1 | 1 | 3 | 0 | 0 | 4 | 1 | 1 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT04426890/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-03): https://cdn.clinicaltrials.gov/large-docs/90/NCT04426890/SAP_001.pdf